CLINICAL TRIAL: NCT04675749
Title: Quality of Life in Female Carriers of X-linked Adrenoleukodystrophy
Brief Title: Quality of Life in Women with X-linked Adrenoleukodystrophy
Acronym: X-ALD_QoL
Status: Recruiting | Type: Observational
Sponsor: Leipzig University Medical Center (Other)
Responsible Party: Principal Investigator, Lisa Schäfer, Dr., Leipzig University Medical Center
Other Study IDs: X-ALD_QoL
Record Dates: First submitted 2020-12-11; First posted 2020-12-19 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: X-linked Adrenoleukodystrophy
Keywords: Adrenoleukodystrophy; Adrenomyeloneuropathy; Brain Diseases, Metabolic, Inborn; Central Nervous System Diseases; Demyelinating Diseases; White Matter Disorder; Genetic Diseases, X-Linked; Peroxisomal Disorders; Metabolic Diseases; Female Carrier; Adrenoleukodystrophy, women; Heterozygous Carrier; Quality of Life
MeSH Terms: conditions — Adrenoleukodystrophy; Brain Diseases, Metabolic, Inborn; Central Nervous System Diseases; Demyelinating Diseases; Genetic Diseases, X-Linked; Peroxisomal Disorders; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
X-linked adrenoleukodystrophy (X-ALD) is a hereditary white matter disorder caused by mutations in the ABCD1 gene leading to disturbances in the metabolism of fatty acids. This results in an accumulation of very long chain fatty acids (VLCFA) in the cells of the body causing damage to the central nervous system (white matter of the brain and spinal cord). The most common adult-onset X-ALD phenotype is adrenomyeloneuropathy (AMN), a slowly progressive myelopathic variant with demyelination of the long tracts in the spinal cord, clinically manifested as slowly progressive spastic paraparesis, sensory ataxia, bladder and sexual dysfunction.

Although this rare disease is inherited X-linked, previous research revealed that up to 80% of heterozygous women develop AMN symptoms during their lifetime.

The primary objectives of this study are 1) to assess the prevalence of symptomatic courses in female carriers of X-ALD and 2) to determine the impact of AMN symptoms on the quality of life of affected women in various areas (including everyday life, work, social network, sleep quality, sexuality, mood).

Participants are asked to fill in self-report questionnaires, which are available in English, German, French, Spanish, and Italian, and are provided electronically on the online platform Leuconnect (https://www.leuconnect.com) launched by European Leukodystrophies Association (ELA) international (https://elainternational.eu/).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from the participant
* Females ≥18 years at the time of consent, with proven X-ALD as defined by

  1. Elevated VLCFA values, or
  2. Mutation in ABCD1 gene

Exclusion Criteria:

* No informed consent and assent
* Current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female carriers of X-ALD with or without AMN symptoms aged ≥18 years
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with AMN Symptoms as Assessed by Adult ALD Clinical Score (AACS) - self-report version | Day 0
Quality of Life in Symptomatic versus Asymptomatic Participants as Assessed by Self-report Questionnaire (SF-36) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Köhler, MD, Principal Investigator — Leipzig University Medical Center, Leukodystrophy Outpatient Clinic, Department of Neurology, Leipzig, Germany
Locations (1):
- Leipzig University Medical Center, Leukodystrophy Outpatient Clinic, Department of Neurology, Leipzig, Germany, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No